CLINICAL TRIAL: NCT03691584
Title: A Phase 1, Open-label, Randomized, PK and Safety Study To Assess Bronchopulmonary Disposition of Intravenous TP-6076 in Healthy Men and Women
Brief Title: Phase 1, Safety and Bronchopulmonary PK Study in Healthy Volunteers
Acronym: BAL
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tetraphase Pharmaceuticals, Inc (Industry)
Collaborators: PRA Health Sciences (Industry)
Responsible Party: Sponsor
Organization: La Jolla Pharmaceutical Company (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: TP-6076-003
Record Dates: First submitted 2018-09-27; First posted 2018-10-02 (Actual); Last update posted 2021-12-17 (Actual); Status verified 2021-12

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — Bronchoalveolar Lavage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BAL PK study (Experimental): Bronchoalveolar lavage procedure performed at either 2, 4, 8, or 24 hours after final dose of TP-6076 on Day 4
  Interventions: Drug: TP-6076; Procedure: Bronchoalveolar lavage

INTERVENTIONS:
Drug: TP-6076 — The dose planned to be administered in this study is an iv infusion of 30 mg TP 6076 q24h for 4 consecutive days (starting on Day 1 and ending on Day 4).
Procedure: Bronchoalveolar lavage — Subjects will be randomized to undergo a BAL at a single time point: either 2, 4, 8, or 24 hours after the start of the final TP-6076 iv infusion on Day 4.
  Other Names: BAL

SUMMARY:
This is a Phase 1, open-label, randomized, PK and safety study in a maximum of 25 healthy subjects who have provided a bronchoalveolar lavage (BAL) sample.

DETAILED DESCRIPTION:
This is a Phase 1, open-label, randomized, PK and safety study in a maximum of 25 healthy subjects who have provided a bronchoalveolar lavage (BAL) sample. The dose planned to be administered in this study is an iv infusion of 30 mg TP 6076 q24h for 4 consecutive days (starting on Day 1 and ending on Day 4).

Subjects will be randomized to undergo a BAL at a single time point: either 2, 4, 8, or 24 hours after the start of the final TP-6076 iv infusion on Day 4. The BAL will be conducted in 5 different subjects at each of the 4 time points, adding up to a total of 20 subjects.

ELIGIBILITY:
Inclusion Criteria:

* The following inclusion criteria must be met for a subject to be eligible for inclusion in the study:

  1. Status : Healthy subject
  2. Gender : Male or female
  3. Age : 18 to 50 years, inclusive, at screening
  4. Body mass index (BMI) : 18.0 to 30.0 kg/m2, inclusive, at screening
  5. Weight : 50 to 105 kg, inclusive, at screening
  6. At screening, females must be non-pregnant and non-lactating, or of non childbearing potential (either surgically sterilized or physiologically incapable of becoming pregnant, or at least 1 year post menopausal [amenorrhoea duration of 12 consecutive months]); non-pregnancy will be confirmed for all females by a serum pregnancy test conducted at screening, admission to the CPU, and follow up.
  7. Post-menopausal females using hormone replacement therapy should be on a stable regimen and be using this since at least 3 months prior to the first study drug administration.
  8. Female subjects of childbearing potential who have a fertile male sexual partner must agree to use adequate contraception from screening until 90 days after the follow up visit. Adequate contraception will be methods with low user dependency (ie, implanted hormonal contraception, an intrauterine device, an intrauterine hormone releasing system, bilateral tubal occlusion, and/or a sole vasectomised male partner with medical assessment). Also, total abstinence, in accordance with the lifestyle of the subject, is acceptable.
  9. Male subjects, if not surgically sterilized, must agree to use adequate contraception when engaging in sexual activity with a female of childbearing potential and not to donate sperm from admission to the CPU until 90 days after the follow-up visit. Adequate contraception for the male subject (and his female partner) will be methods with low user dependency (ie, implanted hormonal contraception, an intrauterine device, an intrauterine hormone releasing system, bilateral tubal occlusion, and/or a sole vasectomised male subject with medical assessment). Also, total abstinence, in accordance with the lifestyle of the subject, is acceptable.
  10. All prescribed medication must have been stopped at least 30 days prior to admission to the CPU. An exception is made for hormonal contraceptives and a stable regimen of hormone replacement therapy, which may be used throughout the study.
  11. All over-the-counter medication, vitamin preparations and other food supplements, or herbal medications (eg, St. John's Wort) must have been stopped at least 14 days prior to admission to the CPU. An exception is made for paracetamol, which is allowed up to admission to the CPU.
  12. Ability and willingness to abstain from alcohol, methylxanthine-containing beverages or food (coffee, tea, cola, chocolate, energy drinks), and grapefruit (juice) from 48 hours prior to admission to the CPU.
  13. Good physical and mental health on the basis of medical history, physical examination, clinical laboratory, ECG, and vital signs, as judged by the Investigator.
  14. Willing to comply with the study procedures.
  15. Willing and able to sign the ICF.

      Exclusion Criteria:

      A subject who meets any of the following exclusion criteria will not be eligible for inclusion in the study:

  <!-- -->

  1. Previous participation in the current study.
  2. Employee of PRA Health Sciences (PRA), Hammersmith Medicines Research Ltd. (HMR), or Tetraphase Pharmaceuticals, Inc.
  3. Subjects who may not tolerate a BAL, or cannot undergo a BAL due to the presence of contraindications to a BAL (including abnormal blood coagulation parameters, refractory hypoxemia, reactive airway disease or asthma, unstable angina or acute myocardial infarction in the 6 months prior to the first study drug administration).
  4. History of any relevant lung disease.
  5. History of relevant drug (including tetracycline-class antibiotics) and/or food allergies.
  6. Using tobacco products or electronic cigarettes within 6 months prior to the first study drug administration.
  7. History of alcohol abuse or drug addiction (including soft drugs like cannabis products) within 2 years prior to the first study drug administration.
  8. Positive drug and alcohol screen (opiates, methadone, cocaine, amphetamines [including ecstasy], cannabinoids, barbiturates, benzodiazepines, tricyclic antidepressants, cotinine, and alcohol) at screening and admission to the CPU.
  9. Average intake of more than 24 units of alcohol per week: 1 unit of alcohol equals approximately 250 mL of beer, 100 mL of wine, or 35 mL of spirits).
  10. Positive screen for hepatitis B surface antigen (HBsAg), antihepatitis C virus (HCV) antibodies, or antihuman immunodeficiency virus (HIV) 1 and 2 antibodies.
  11. Participation in a drug study within 60 days prior to the first study drug administration in the current study. Participation in more than 3 other drug studies in the 10 months prior to the first study drug administration in the current study.
  12. Donation or loss of more than 400 mL of blood within 90 days prior to the first study drug administration. Donation or loss of more than 1.5 liters of blood (for male subjects)/more than 1.0 liters of blood (for female subjects) in the 10 months prior to the first study drug administration in the current study.
  13. Significant and/or acute illness within 5 days prior to the first study drug administration that may impact safety assessments, in the opinion of the Investigator.
  14. Unsuitable veins for infusion or blood sampling.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2018-11-26 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-12-18 (Actual)

PRIMARY OUTCOMES:
Concentrations of TP-6076 in plasma | Up to 2, 4, 8, or 24 hours after the start of the final TP-6076 iv infusion on Day 4.
  Pharmacokinetics
Concentrations of TP-6076 in epithelial lining fluid (ELF) | Up to 2, 4, 8, or 24 hours after the start of the final TP-6076 iv infusion on Day 4.
Concentrations of TP-6076 in alveolar macrophages (AMs) | Up to 2, 4, 8, or 24 hours after the start of the final TP-6076 iv infusion on Day 4.
maximum observed concentration (Cmax) | Up to 2, 4, 8, or 24 hours after the start of the final TP-6076 iv infusion on Day 4.
time to maximum observed concentration (Tmax) | Up to 2, 4, 8, or 24 hours after the start of the final TP-6076 iv infusion on Day 4.

SECONDARY OUTCOMES:
collection of adverse events | Screening through Day 20 (+/- 5 days)

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Dennison, MD, Principal Investigator — Hammersmith Medicines Research
Locations (1):
- Hammersmith Medicines Research, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No